CLINICAL TRIAL: NCT02216409
Title: A First-in-Human Phase 1 Dose Escalation Trial of Hu5F9-G4 in Patients With Advanced Solid Malignancies
Brief Title: Phase 1 Trial of Hu5F9-G4, a CD47-targeting Antibody
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCI-CD47-001
Record Dates: First submitted 2014-08-12; First posted 2014-08-15 (Estimated); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Solid Tumor
MeSH Terms: interventions — magrolimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Hu5F9-G4) (Experimental): Hu5F9-G4 monotherapy
  Interventions: Drug: Hu5F9-G4

INTERVENTIONS:
Drug: Hu5F9-G4

SUMMARY:
The purpose of this study is to assess the safety and tolerability of Hu5F9-G4 in participants with solid tumors.

DETAILED DESCRIPTION:
This is a first-in-human, first-in-class, escalating dose trial of an antibody that inhibits an anti-apoptotic signal in human macrophages. The major aims of the study are to define the safety profile of this new drug, and to determine a recommended dose and schedule for potential additional trials.

ELIGIBILITY:
Inclusion Criteria:

Patients with histologically or cytologically confirmed advanced solid malignancy or Lymphoma

Relapsed or refractory disease after at least 1 prior systemic treatment for the primary malignancy and not a candidate for other curative treatment.

Adequate hematologic status

Adequate coagulation function

Adequate hepatic function

Adequate renal function

Exclusion Criteria:

Known primary tumors of central nervous system disease

Known active brain metastases

Known cardiopulmonary disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of Hu5F9-G4 | The first 28 days on study, for determination of Dose Limiting Toxicities
  The CTCAE criteria will be used to assess adverse events on this trial.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Takimoto, MD, Study Chair — Gilead Sciences
Locations (6):
- United States (6):
  - Stanford Cancer Institute, Stanford, California
  - University of Chicago, Chicago, Illinois
  - START Midwest, Grand Rapids, Michigan
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Oklahoma, Oklahoma City, Oklahoma
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas

REFERENCES:
- [Derived] Sikic BI, Lakhani N, Patnaik A, Shah SA, Chandana SR, Rasco D, Colevas AD, O'Rourke T, Narayanan S, Papadopoulos K, Fisher GA, Villalobos V, Prohaska SS, Howard M, Beeram M, Chao MP, Agoram B, Chen JY, Huang J, Axt M, Liu J, Volkmer JP, Majeti R, Weissman IL, Takimoto CH, Supan D, Wakelee HA, Aoki R, Pegram MD, Padda SK. First-in-Human, First-in-Class Phase I Trial of the Anti-CD47 Antibody Hu5F9-G4 in Patients With Advanced Cancers. J Clin Oncol. 2019 Apr 20;37(12):946-953. doi: 10.1200/JCO.18.02018. Epub 2019 Feb 27. PMID 30811285
- [Derived] Liu J, Wang L, Zhao F, Tseng S, Narayanan C, Shura L, Willingham S, Howard M, Prohaska S, Volkmer J, Chao M, Weissman IL, Majeti R. Pre-Clinical Development of a Humanized Anti-CD47 Antibody with Anti-Cancer Therapeutic Potential. PLoS One. 2015 Sep 21;10(9):e0137345. doi: 10.1371/journal.pone.0137345. eCollection 2015. PMID 26390038